CLINICAL TRIAL: NCT04411680
Title: A Phase 2 Trial Evaluating Sargramostim in Patients With COVID-19 Associated Acute Hypoxemia
Brief Title: Study of Sargramostim in Patients With COVID-19
Acronym: iLeukPulm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Partner Therapeutics, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTX-001-002
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Results first posted 2022-02-18 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: COVID-19; sargramostim; Leukine; rhu-GM-CSF; acute hypoxemia; iLeukPulm; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Standard of Care

STUDY DESIGN:
Intervention Model Description: This Phase 2, randomized, open-label study will enroll approximately 120 patients with COVID-19 associated acute hypoxemia. It is a randomized 2:1 study to evaluate sargramostim treatment plus institutional standard of care compared to institutional standard of care alone.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sargramostim Arm (Experimental): Day 1 - 5: Sargramostim treatment in addition to standard of care for COVID-19
  Interventions: Drug: Sargramostim; Drug: Standard of care
- Control Arm (Active Comparator): Standard of care for COVID-19
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Sargramostim — Sargramostim is a glycosylated, yeast-derived recombinant human granulocyte-macrophage colony stimulating factor (rhu-GM-CSF). Dosage for inhaled sargramostim: 125 mcg twice a day. Dosage for intravenous sargramostim: 125mcg/m2/day given over a 4 hour period.
  Other Names: Leukine; GM-CSF
  Arms: Sargramostim Arm
Drug: Standard of care — Standard of care for COVID-19

SUMMARY:
The purpose of this research is to find out if a drug (sargramostim) also known as Leukine® could help patient recover faster from COVID-19. Sargramostim may help the lungs recover from the effects of COVID-19, and this research study will help to find this out.

DETAILED DESCRIPTION:
This Phase 2 study is designed as a proof of concept study and will randomize 2:1 approximately 120 patients with COVID-19 associated acute hypoxemia: of which 80 patients will receive sargramostim plus standard of care, and 40 patients who will receive standard of care alone. The aim of the study is to determine if inhaled sargramostim, as an adjunct to institutional standard of care, improves clinical outcomes in patients with COVID-19-associated acute hypoxemia. All patients on the sargramostim arm will be treated with 125 mcg inhaled sargramostim twice daily for 5 days, in addition to institutional standard of care. If required, upon progression to an invasive mechanical ventilator, administration of sargramostim may be delivered by intravenous infusion to complete a total of 5 days (including days delivered via inhalation).

GM-CSF is a critical cytokine for healthy pulmonary function and is necessary for the maturation and maintenance of alveolar macrophages. Preclinical studies have shown GM-CSF confers resistance to influenza by enhancing innate immune mechanisms that depend on alveolar macrophages for their health and normal functioning. Clinical studies of sargramostim in patients with severe sepsis and respiratory dysfunction or acute respiratory distress syndrome have shown improvements in oxygenation and lung compliance.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients (or legally authorized decision maker) must provide informed consent
* Test positive for SARS-CoV-2 virus by PCR
* Admitted to hospital
* Presence of acute hypoxemia defined as (either or both)

  * saturation below 93% on ≥ 2 L/min oxygen supplementation
  * PaO2/FiO2 below 350

Exclusion Criteria:

* Patients requiring invasive (mechanical ventilation) or non-invasive (CPAP, BiPAP for hypoxemia) ventilation or ECMO (Note: oxygen supplementation using high flow oxygen systems or low flow oxygen systems would not exclude patients from this study)
* Intractable metabolic acidosis
* Cardiogenic pulmonary edema
* Hypotension requiring use of vasopressors
* Hyperferritinemia (serum ferritin ≥2,000 mcg/L)
* White blood cell count > 50,000/mm3
* Participation in another interventional clinical trial for COVID-19 therapy
* Highly immunosuppressive therapy or anti-cancer combination chemotherapy within 24 hours prior to first dose of sargramostim
* Known or suspected intolerance or hypersensitivity to sargramostim, or any component of the product
* Previous experience of severe and unexplained side effects during aerosol delivery of any kind of medical product
* Presence of any preexisting illness that, in the opinion of the Investigator, would place the patient at an unreasonably increased risk through participation in this study
* Pregnant or breastfeeding females
* Severe or uncontrolled pulmonary comorbid conditions, including systemic steroid dependent asthma, systemic steroid dependent COPD, oxygen dependent COPD, lung transplant, known interstitial lung disease, or cystic fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Information, Study Director — Partner Therapeutics, Inc.
Locations (11):
- United States (11):
  - St. Jude Medical Center, Fullerton, California
  - St. Joseph Hospital of Orange, Orange, California
  - California Pacific Medical Center - Van Ness Campus, San Francisco, California
  - TidalHealth Peninsula Regional, Inc, Salisbury, Maryland
  - University of Missouri Health Care, Columbia, Missouri
  - Great Plains Health, North Platte, Nebraska
  - Richmond University Medical Center, Staten Island, New York
  - Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - University of Toledo Medical Center, Toledo, Ohio
  - Memorial Hermann Hospital Affiliated with the University of Texas Health Science Center at Houston, McGovern Medical School, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paine R, Chasse R, Halstead ES, Nfonoyim J, Park DJ, Byun T, Patel B, Molina-Pallete G, Harris ES, Garner F, Simms L, Ahuja S, McManus JL, Roychowdhury DF. Inhaled Sargramostim (Recombinant Human Granulocyte-Macrophage Colony-Stimulating Factor) for COVID-19-Associated Acute Hypoxemia: Results of the Phase 2, Randomized, Open-Label Trial (iLeukPulm). Mil Med. 2023 Jul 22;188(7-8):e2629-e2638. doi: 10.1093/milmed/usac362. PMID 36458916

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was randomized to the sargramostim arm and then withdrew consent prior to treatment.
Groups:
- Sargramostim Arm: Day 1 - 5: Sargramostim treatment in addition to standard of care for COVID-19
  Sargramostim: Sargramostim is a recombinant human granulocyte-macrophage colony stimulating factor (rhu-GM-CSF). Dosage for inhaled sargramostim: 125 mcg twice a day. Dosage for intravenous sargramostim: 125mcg/m2/day given over a 4 hour period.
  Standard of care: Standard of care for COVID-19
Period: Treatment Period
Arm/Group | Sargramostim Arm | Control Arm
Started | 78 | 44
Completed | 49 | 36
Not Completed | 29 | 8
Not completed — Adverse Event | 3 | 0
Not completed — Discharged from hospital | 18 | 7
Not completed — Missed 1 or more doses | 8 | 0
Not completed — Transferred to another hospital | 0 | 1
Period: Follow up Period
Arm/Group | Sargramostim Arm | Control Arm
Started | 78 | 44
Completed | 60 | 30
Not Completed | 18 | 14
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 5 | 6
Not completed — Death | 11 | 8

BASELINE CHARACTERISTICS:
Population: One patient was randomized to the Sargramostim Arm, but was not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sargramostim Arm | Control Arm | Total
Number analyzed (Participants) | 78 | 44 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 30 | 77
  >=65 years | 31 | 14 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (13.00) | 58.2 (10.61) | 60.4 (12.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 18 | 61
  Male | 35 | 26 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 11 | 35
  Not Hispanic or Latino | 53 | 33 | 86
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 6 | 1 | 7
  White | 48 | 33 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 20 | 9 | 29
Body Mass Index [Mean (Standard Deviation); unit: kilograms/meter squared] — Population: Data to calculate BMI is missing for 5 patients in sargramostim arm and 1 patient in control arm.
  kilograms/meter squared
    number analyzed (Participants) | 73 | 43 | 116
    (all) | 34.86 (8.988) | 35.44 (9.647) | 35.07 (9.200)

OUTCOME MEASURES:

1. Primary Outcome: Change in Oxygenation Parameter of P(A-a)O2 Gradient by Day 6
Description: The P(A-a)O2 gradient is a measure of how well the oxygen moves from the lungs into the bloodstream. Patients with a high gradient have less oxygen in the bloodstream.
Time Frame: 1-6 days
Population: Patients analyzed if they had both a baseline and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | Sargramostim Arm | Control Arm
Number analyzed (Participants) | 63 | 33
millimeters of mercury (mmHg) | -102.3 (19.44) | -30.5 (26.88)

2. Primary Outcome: Number of Patients Who Have Been Intubated by Day 14
Time Frame: 1-14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sargramostim Arm | Control Arm
Number analyzed (Participants) | 78 | 44
Participants | 9 | 7

3. Secondary Outcome: Change in Ordinal Scale
Description: The ordinal scale was used, where 0 is not hospitalized, no clinical or virological evidence of infection, and 8 is death.
Time Frame: 1-28 days
Population: Only 86 patients had follow up data at Day 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sargramostim Arm | Control Arm
Number analyzed (Participants) | 61 | 25
score on a scale | -2.6 (1.49) | -2.5 (1.48)

4. Secondary Outcome: All Cause 28-day Mortality
Time Frame: 1-28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sargramostim Arm | Control Arm
Number analyzed (Participants) | 78 | 44
Participants | 9 | 6

5. Secondary Outcome: Number of Patients With Treatment-related Adverse Events
Description: Number of patients with side effects related to treatment with sargramostim. Patients on the control arm did not receive sargramostim.
Time Frame: 1-58 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sargramostim Arm | Control Arm
Number analyzed (Participants) | 78 | 44
Participants | 5 | 0

6. Secondary Outcome: Survival Time of Patients
Time Frame: Day 1-90
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sargramostim Arm | Control Arm
Number analyzed (Participants) | 78 | 44
Days | 76.0 (27.05) | 72.6 (28.56)

7. Secondary Outcome: Causes of Death
Time Frame: Day 1-90
Population: Patients alive at Day 90 were not analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Sargramostim Arm | Control Arm
Number analyzed (Participants) | 11 | 8
Participants
  Acute respiratory distress syndrome | 4 | 2
  Respiratory failure | 6 | 3
  Cardiorespiratory arrest | 1 | 2
  Septic shock | 0 | 1

8. Secondary Outcome: Change From Baseline in P/F Ratio
Description: The P/F ratio is a simple way to assess severity of low blood oxygen. It's the ratio of PaO2 (arterial oxygen partial pressure obtained from an arterial blood gas) to FiO2 (fraction of inspired oxygen expressed as a decimal). A normal arterial blood is gas 80 to 100 mm Hg. Normal room air has 21% or 0.21 oxygen. So a "normal" P/F ratio is about 380-475. A high P/F ratio means more oxygen in the bloodstream and a low P/F ratio means less oxygen in the bloodstream.
  This outcome measure compares the improvement (increase) in P/F ratio between treatment arms.
Time Frame: From Day 1 up to Day 6
Population: Patients were analyzed if they had both a baseline and at least 1 post-baseline measurement of P/F ratio.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sargramostim Arm | Control Arm
Number analyzed (Participants) | 63 | 33
ratio | 65.70 (97.964) | 47.24 (99.942)

9. Secondary Outcome: Number of Participants Wtih Nosocomial Infections
Description: Nosocomial infections also referred to as healthcare-associated infections (HAI), are infection(s) acquired during the process of receiving health care that was not present during the time of admission.
Time Frame: Day 1-90
Measure: Count of Participants; unit: Participants
Arm/Group | Sargramostim Arm | Control Arm
Number analyzed (Participants) | 78 | 44
Participants | 0 | 0

10. Secondary Outcome: Number of Patients Requiring Invasive Mechanical Ventilation
Description: The is the number of patients that needed to be placed on a ventilator.
Time Frame: Day 1-90
Measure: Count of Participants; unit: Participants
Arm/Group | Sargramostim Arm | Control Arm
Number analyzed (Participants) | 78 | 44
Participants | 12 | 9

11. Secondary Outcome: Duration of Invasive, Non-invasive and Supplemental Oxygen
Description: This endpoint includes duration of any/all types of respiratory support
Time Frame: Day 1-90
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sargramostim Arm | Control Arm
Number analyzed (Participants) | 78 | 44
Days | 37.9 (35.64) | 32.8 (34.25)

12. Secondary Outcome: Duration of Hospitalization
Time Frame: Day 1-90
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sargramostim Arm | Control Arm
Number analyzed (Participants) | 78 | 44
Days | 12.1 (9.39) | 11.8 (8.63)

13. Secondary Outcome: Time to Normalization of White Blood Cells and Lymphocytes
Description: Normalization of WBC and lymphocyte count is defined as whether WBC and lymphocyte count results are normal or below normal or above normal ranges at available visits.
Time Frame: Day 1-90
Population: Of 78 and 44 participants in the Sargramostim and Control Arms, respectively, only 28 (35.8%) and 17 (38.6%) had both baseline and post-baseline values available for evaluation at the Day 6 timepoint of interest.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sargramostim Arm | Control Arm
Number analyzed (Participants) | 28 | 17
Days | NA (NA) — Insufficient number of participants with events | NA (NA) — Insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: Adverse Events: Day 1-58, All-Cause Mortality: Day 1-90
Arm/Group | Sargramostim Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 11/78 | 8/44
Serious Adverse Events (participants affected / at risk) | 15/78 | 14/44
Other Adverse Events (participants affected / at risk) | 47/78 | 30/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sargramostim Arm (N=78) | Control Arm (N=44)
Atrial fibrillation (Cardiac disorders) | 1 | 1 — Abnormal heartbeat
Atrial flutter (Cardiac disorders) | 0 | 1 — Abnormal heartbeat
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiac death (General disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 — Skin infection
Septic shock (Infections and infestations) | 0 | 2 — Shock due to infection
False positive investigation result (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 — Too much potassium in the blood stream
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Anuria (Renal and urinary disorders) | 0 | 1 — Absence of urination
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Emphysema
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Not enough oxygen in the bloodstream
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 — Blood clot in the lungs
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 5 — Term respiratory failure includes terms respiratory failure, acute respiratory failure and chronic respiratory failure
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sargramostim Arm (N=78) | Control Arm (N=44)
Anemia (Blood and lymphatic system disorders) | 5 | 3 — Not enough red blood cells
Constipation (Gastrointestinal disorders) | 7 | 3
Septic shock (Infections and infestations) | 5 | 1 — Shock due to infection
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 4 — Too much glucose in the bloodstream
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 3 — Too little potassium in the bloodstream
Anxiety (Psychiatric disorders) | 4 | 4
Insomnia (Psychiatric disorders) | 3 | 4
Acute kidney injury (Renal and urinary disorders) | 3 | 4
Hypotension (Vascular disorders) | 5 | 4 — Low blood pressure

LIMITATIONS AND CAVEATS:
Limitations include lack of a blinded placebo control and reliance on ABG measurement for estimation of P(A-a)O2 gradient. Some clinical endpoints trial might have been affected by observer bias, availability of hospital or ICU resources, and/or hospital discharge. Missing ABG measurements may have resulted from decreased standard utilization of ABG in recent years, and hospital staff overload due to the COVID-19 pandemic may have led to absent follow-up assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT04411680/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT04411680/SAP_001.pdf